CLINICAL TRIAL: NCT04146675
Title: Pilot Study for the Evaluation of a T-shirt "Balance" Containing Ceramic Fibers
Brief Title: Evaluation of a T-shirt "Balance" Containing Ceramic Fibers
Acronym: Equi-tee-shirt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2013_06; 2013-A00727-38 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2019-01-09; First posted 2019-10-31 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-01

CONDITIONS: Geriatrics
Keywords: Gerontology; elderly,; falls; balance and walking disorders.

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRICOT JERSEY VANISE DOUBLE FACE (Experimental)
  Interventions: Device: TRICOT JERSEY VANISE DOUBLE FACE
- TRICOT JERSEY SIMPLE (Placebo Comparator)
  Interventions: Device: TRICOT JERSEY SIMPLE

INTERVENTIONS:
Device: TRICOT JERSEY VANISE DOUBLE FACE — Short sleeve t-shirt : TRICOT JERSEY VANISE DOUBLE FACE " THERMOLACTYL EVOLUTION " with ceramic fibers.
  A Tinetti test will be performed while wearing the T-shirt, as well as an evaluation of the equilibration on posturography platform under static conditions and an assessment of dynamic equilibrium and locomotion in motion analysis.
  Arms: TRICOT JERSEY VANISE DOUBLE FACE
Device: TRICOT JERSEY SIMPLE — Short sleeve t-shirt : TRICOT JERSEY SIMPLE The comparator T-shirt has the same weight, the same appearance, and will be used by patients in the same way and under the same conditions as the T-shirt with ceramic fibers.
  Arms: TRICOT JERSEY SIMPLE

SUMMARY:
Falls are frequent and often serious events in the elderly. The consequences of falls are often severe: traumatic (fractures, hematomas, ..) and psychological. Falls are among the top ten causes of death in this population and, for people older than 70, falls are the leading cause of accidental death.

The Damart company has developed a fabric containing ceramic fibers. Clothes containing such fibers have been found to improve balance.

This study aims to measure the effect of a t-shirt with a ceramic membrane ("ceramic" t-shirt) on the balance and walking compared to the effect of a "placebo" t-shirt (same weight, appearance and texture).

The hypothesis is that wearing the ceramic tee-shirt significantly improves balance and walking, suggesting that it can also reduce falls - the main consequence of the balance and walking disorder.

ELIGIBILITY:
Inclusion Criteria:

* Presenting disturbances of balance (determined by a Tinetti test score strictly greater than 12)
* Hold the balance while standing with his feet and arms along the body and walk for 3 meters without major imbalance that may cause a fall
* Consent to participate in the study (a signed written consent form)
* Covered by a social security system

Exclusion Criteria:

* A motor deficit of the lower limbs focused and characterized by neurological or orthopedic cause (for example hemiplegia after a cerebrovascular accident, limb amputation).
* Inability to receive the protocol information
* Inability to participate in the entire study
* Absence of a social security coverage
* Refusal to sign the Informed Consent form

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Variation of the Tinetti score between the two group | Baseline
  Variation of the Tinetti score between the group T-shirt placebo (Δ Tinetti T-shirt placebo vs Tinetti clothing patients) and the ceramic tee-shirt group (Δ Tinetti ceramic t-shirt vs Tinetti clothing patients).
  Scoring of the Tinetti Assessment Tool is done on a three point ordinal scale with a range of 0 to 2.
  A score of 0 represents the most impairment, while a score of 2 represents independence. The individual scores are then combined to form three measures; an overall gait assessment score, and overall balance assessment score, ad a combined gait and balance score.

SECONDARY OUTCOMES:
variation of the posturography technique | Baseline
  Parameters of the static equilibrium produced by the posturography technique: the length of the balancing path (mm)
variation of motion analysis (the optoelectronic system (VICON®) | Baseline
  Parameters of the dynamic equilibrium and locomotion produced by the technique of motion analysis.
  Analysis of gait parameters: speed (seconde) and length (meters). these parameters will be combined to report the dynamic equilibrium and locomotion

CONTACTS AND LOCATIONS:
Overall Officials: François Puisieux, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital gériatrique les Bateliers, Lille, France

IPD SHARING:
Plan to Share IPD: Undecided